CLINICAL TRIAL: NCT01901588
Title: Efficacy of Single-Shot Dexmedetomidine Versus Placebo in Preventing Pediatric Emergence Delirium in Strabismus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S12-00556
Record Dates: First submitted 2013-04-17; First posted 2013-07-17 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Strabismus; Delirium on Emergence; Pediatric Disorders
Keywords: strabismus; pediatric; emergence delirium; precedex/dexmedetomidine
MeSH Terms: conditions — Strabismus; Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): dexmedetomidine/precedex
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): patients receive saline solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dose of dexmedetomidine 0.3 mcg/kg over 5 minutes
  Other Names: Precedex
  Arms: Dexmedetomidine
Other: Placebo — intraoperative dose of intravenous placebo
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
This study is trying to see if using precedex pre-operatively prevents emergence delirium in pediatric (ages 1-7) patients undergoing strabismus surgery.

DETAILED DESCRIPTION:
Emergence delirium (ED) is a complex behavioral disturbance characterized by psychomotor agitation, perceptual disturbances, delusions, and disorientation during recovery from general anesthesia. In the population of subjects who undergo strabismus surgery, there are multiple factors that may increase the risk of ED. These include age, typically preschool children aged 1-7 years, rapid surgical times with rapid awakening, use of sevoflurane as the primary anesthetic, and surgically-induced postoperative visual disturbance. The aims of this study are: 1) To examine whether post-induction treatment with an α-2 receptor agonist, precedex (dexmedetomidine), decreases postoperative emergence agitation after strabismus surgery compared to placebo, and 2) to determine whether treatment has any effect on postoperative pain, nausea/vomiting, number of pain-related interventions, and time to PACU discharge. We hypothesize that precedex will attenuate the ED response greater than placebo or a lower dose after strabismus surgery and will reduce PACU pain scores without increasing PACU length of stay.

Inclusion:

i. Pediatric patients aged 1-7 years of age ii. American Society of Anesthesiologists (ASA) physical status I-II iii. No significant laboratory abnormalities

Exclusion:

i. Presence of medicated behavioral disorder ii. Subjects for which precedex, opiates, benzodiazepines, or inhalational anesthetics are contraindicated iii. Parental refusal

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status of I or II
* male or female, aged 1-7
* has no significant lab abnormalities

Exclusion Criteria:

* ASA physical status of III, IV or V
* Presence of medicated behavioral disorder
* Subjects for which dexmedetomidine, opiates, benzodiazepines or inhalational anesthetics are contraindicated.
* Parental refusal

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Brown, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient's familes were approached on the day of surgery and spoken to privately in the pre-op area. Fliers were placed at the phthalmalogist's offices so were generally aware of the study ahead of time.
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 31 | 63
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 20 | 15 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan | 0 | 0 | 0
  Asian or Pacific Islander | 1 | 2 | 3
  Black, Not of Hispanic-American Origin | 2 | 1 | 3
  Hispanic-American | 1 | 0 | 1
  White, not of Hispanic-American Origin | 23 | 22 | 45
  Other or Unknown | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Pediatric Emergence Delirium in Strabismus Surgery
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
percentage of participants | 50 | 48

2. Secondary Outcome: Percentage of Participants Receiving Pain Medication
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
percentage of participants | 50 | 66

3. Secondary Outcome: Post-op Pain Interventions
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Number; unit: number of pain interventions/group
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
number of pain interventions/group | 18 | 30

4. Secondary Outcome: Percentage of Participants Requiring Post-operative Nausea and Vomiting (PONV) Rescue Medications
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Number; unit: percentage of participants
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
percentage of participants | 0 | 14

5. Secondary Outcome: Time to Arousal
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
minutes | 60 (36) | 40 (39)

6. Secondary Outcome: Time to PACU Discharge
Time Frame: Length of PACU stay (around 3 hours on average)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 26 | 29
minutes | 186 (64) | 173 (60)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes